CLINICAL TRIAL: NCT04311580
Title: Intravesical Electromotive Mitomycin for High Risk Urothelial Non-muscle Invasive Bladder Cancer After Intravesical Bacillus Calmette-Guérin Failure
Brief Title: Intravesical Electromotive Mitomycin After Bacillus Calmette-Guérin Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rome Tor Vergata (Other)
Collaborators: University of Bari (Other)
Responsible Party: Principal Investigator, Savino Mauro Di Stasi, ASSOCIATE PROFESSOR OF UROLOGY, University of Rome Tor Vergata
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UTV/08-05-95
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Bladder Cancer
Keywords: non-muscle invasive bladder cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- urothelial high risk non-muscle invasive bladder cancer (Experimental): patients with urothelial high risk non-muscle invasive bladder cancer after failed intravesical bacillus Calmette-Guérin treatment.
  Interventions: Combination Product: intravesical electromotive administration of mitomycin

INTERVENTIONS:
Combination Product: intravesical electromotive administration of mitomycin

SUMMARY:
Patients with urothelial high risk non-muscle invasive bladder cancer patients will be treated with intravesical electromotive drug administration/mitomycin (EMDA/MMC) after bacillus Calmette-Guerin (BCG) failure. Patients are scheduled for an initial 6 weekly treatments, a further 6 weekly treatments for non-responders and a followup 10 monthly treatments for responders. Complete response will be defined as histological disappearance of malignancy on bladder biopsy and resolution of abnormal cytological findings after treatment. Time to first recurrence, time to progression, overall survival, and disease-specific survival wil be estimated by use of the Kaplan-Meier method.

DETAILED DESCRIPTION:
Partecipants

Inclusion criteria:

* Patients with urothelial high risk NMIBC (high grade stage Ta, T1 and/or carcinoma in situ) after intravesical BCG failure;
* adequate bone marrow reserve;
* normal renal function;
* normal liver function;
* Karnofsky performance score of 50 to 100.

Exclusion criteria:

* non-urothelial carcinomas of the bladder;
* known allergy to MMC;
* previous or concomitant urothelial carcinoma of the upper urinary tract and urethra, or both;
* bladder capacity less than 200 mL;
* untreated urinary-tract infection;
* severe systemic infection (ie, sepsis);
* urethral strictures that would prevent endoscopic procedures and catheterisation;
* other concurrent chemotherapy, radiotherapy, and treatment with biological response modifiers;
* other malignant diseases within 5 years of start of EMDA MMC (except for adequately treated basal-cell or squamous-cell skin cancer, in situ cervical cancer);
* pregnancy;
* psychological, familial, sociological, or geographical factors that would preclude study participation.

The institutional review boards of each participating centre approved the study design. all enrolled patients will sign an informed consent form, approved by the institutional review boards, providing details of treatments.

BCG Failure

The definition of BCG failure in patients has been proposed as follows:

1. BCG-refractory disease when there is failure to achieve a disease-free state at 6 months following initial BCG therapy with either maintenance or retreatment at 3 months because of persistent or rapidly recurrent tumor;
2. BCG-resistant disease when there is recurrence or persistence at 3 months following an induction cycle;
3. BCG-relapsing disease when the disease recurs after the patient is disease-free for 6 months;
4. BCG-intolerant disease when the disease recurs following administration of a less than adequate course of therapy because of a serious adverse event or symptomatic intolerance that requires discontinuation of further BCG therapy.13 Study design Patients will underwent: upper urinary tract imaging, urinary cytology of the bladder and upper urinary tract; random cold-cup biopsies of the bladder and prostatic urethra-ie, sampling of seemingly healthy urothelium and of suspicious areas; and complete transurethral resection (TUR) of all bladder tumour visible on endoscopy, ensuring muscle was included in resected samples. All patients will underwent re-staging TUR 4-5 weeks later. All clinical assessors are adequately trained in the above procedures, and no methods are used to enhance the quality of measurements. All biopsy samples of tumour and bladder will be reviewed by a pathologist for stage and grade. Tumour stage are classified according to the 1997 TNM classification of the International Union Against Cancer, and tumour grade was defined in accordance with the 1973 WHO classification.

Treatment schedule All patients will start induction EMDA/MMC of 6 intravesical treatments at weekly intervals commencing 2-3 weeks after re-staging TUR. Intravesical EMDA MMC is given by a battery-powered generator delivering a controlled electric current that passes between the active intravesical electrode integrated into a specific transurethral catheter and dispersive ground electrodes on skin of the lower abdomen (Physion srl, Mirandola, Italy). Patients are placed on fluid restriction and 2 g ingested sodium bicarbonate the night before treatment, the morning of treatment, and 2 h before treatment with mitomycin. The bladder is emptied through the electrode-transurethral-catheter and 40 mg mitomycin dissolved in 100 mL water was infused intravesically by gravity and retained in the bladder for 30 min, while 20 mA for 30 min pulsed electric current was given externally. Two dispersive cathode electrodes were placed on lower abdominal skin that had been degreased with alcohol. The bladder was then emptied and the catheter removed.

Patients who were disease-free 3 months after treatment were scheduled to receive monthly infusions of BCG for 10 months. Maintenance treatment was given to the same dose and methods of infusion as initial allocated treatment. Response to treatment was assessed with abdominal ultrasonography, cystoscopy, and urinary cytology. In patients who were free of disease 3 months after treatment, these assessments were done every 3 months during the first 3 years and every 6 months thereafter. Patients with carcinoma in situ underwent abdominal ultrasonography, cystoscopy, urinary cytology, and random bladder biopsies at 3 months and 6 months. If bladder cytology was positive for cancer cells but no lesions were visible on cystoscopy, cytology of the upper urinary tract and random biopsies of the bladder and prostatic urethra were done. If, at 3 months' follow-up, carcinoma in situ persisted or a superficial tumour recurred (ie, stage pTa tumour confined to the urothelium or stage pT1 with invasion of the lamina propria), the patient underwent multiple, random biopsy sampling and TUR of all bladder tumour visible on endoscopy and received a second course of intervention treatment.

Cystoscopy, biopsies, and urinary cytology were repeated 3 months after the start of the second course. Patients who were disease-free after the second course of treatment received the full course of monthly maintenance instillations (ie, one infusion of electromotive mitomycin for 10).

Patients were suspended from the trial on a second recurrence, on persistence of carcinoma in situ, on development of carcinoma in the upper-urinary tract or prostatic urethra, on progression to muscle-invasive disease (ie, stage pT2 or more advanced), or on development of metastases. Further treatment was left to the discretion of the local investigator.

Toxicity Side effects were classified as local, systemic or allergic. Local toxicity was defined as culture proven bacterial cystitis, drug induced (chemical) cystitis and other localized effects. Systemic side effects were defined as fever exceeding 38C, general malaise and fatigue. Skin rash was regarded as allergic reaction. The severity of side effects were classified by the treating physician, with subsequent decision to continue, delay or abandon treatment.

Patient follow-up. Response to treatment was assessed with cystoscopy, urinary cytology and /or biopsy only if indicated by suspicious cytological findings or on cystoscopy. In disease-free cases, cystoscopy and urinary cytology were repeated at 3-month intervals for 2 years, 6-month intervals for 3 years and yearly thereafter.

Patient evaluation Patients with stage pTa and pT1 tumour without carcinoma in situ are classified as disease-free and therefore treated prophylactically; those with carcinoma in situ are treated therapeutically, and response is scored as no response or as complete response. Complete response is defined as complete disappearance of carcinoma in situ, as documented by a normal cytology, cystoscopy, and random bladder biopsies.

The primary endpoint is disease-free interval for patients without carcinoma in situ and for patients with carcinoma in situ who are disease-free after treatment-ie, time from enrollment to first cystoscopy noting recurrence. Patients with carcinoma in situ who did not have complete response after 3 months of treatment are regarded as having recurrence with no follow-up. The secondary endpoints are time to progression, overall survival, and disease specific survival. Time to progression is defined as time from randomisation until the onset of muscle invasive disease as recorded by pathological assessment of TUR samples or biopsy samples. Overall survival is defined as time from enrollment until death from any cause; disease specific survival as time from enrollment until death from bladder cancer. Patients without recurrence or progression are censored at the last cystoscopy, and those lost to follow-up were censored at the last known day of survival.

Statistical Analysis All analyses are done by intention to treat. Time to first recurrence, time to progression, overall survival, and disease-specific survival are estimated by use of the Kaplan-Meier method. Comparisons are estimated by use of log-rank test. All tests are two-sided, and p<0·05 was regarded as significant. The investigators will calculated hazard ratios with 95% CI by use of proportional-hazards regression.

ELIGIBILITY:
Inclusion Criteria:

* Patients with urothelial high risk non-muscle invasive bladder cancer (high grade stage Ta, T1 and/or carcinoma in situ) after intravesical BCG failure;
* adequate bone marrow reserve;
* normal renal function;
* normal liver function;
* Karnofsky performance score of 50 to 100;

Exclusion Criteria:

* Non-urothelial carcinomas of the bladder;
* known allergy to mitomicyn ;
* previous or concomitant urothelial carcinoma of the upper urinary tract and urethra, or both;
* bladder capacity less than 200 mL;
* untreated urinary-tract infection; severe systemic infection (ie, sepsis);
* urethral strictures that would prevent endoscopic procedures and catheterisation;
* other concurrent chemotherapy, radiotherapy, and treatment with biological response modifiers;
* other malignant diseases within 5 years of start of EMDA MMC (except for adequately treated basal-cell or squamous-cell skin cancer, in situ cervical cancer);
* pregnancy;
* psychological, familial, sociological, or geographical factors that would preclude study participation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2020-03-10 (Actual)

PRIMARY OUTCOMES:
Time to first recurrence | Up to 100 monthss. Time from enrollment to first cystoscopy noting disease recurrence.
  Time from enrollment to first cystoscopy noting disease recurrence.

SECONDARY OUTCOMES:
Time to disease progression | Up to 100 months. Time from randomisation until the onset of muscle invasive disease
  Time from randomisation until the onset of muscle invasive disease

OTHER OUTCOMES:
Overall survival, and disease-specific survival | Up to 100 months. Time from enrolment until death from any cause; disease specific survival as time from enrollment until death from bladder cancer
  Time from enrolment until death from any cause; disease specific survival as time from enrollment until death from bladder cancer

CONTACTS AND LOCATIONS:
Overall Officials: SAVINO M DI STASI, Principal Investigator — TOR VERGATA UNIVERSITY OF ROME

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: January 2024. Data will become available and for 24 months
Access Criteria: Anyone who wishes to access the data.
URL: http://directory.uniroma2.it/index.php/schede/getCV/4053

REFERENCES:
- [Result] Di Stasi SM, Vespasiani G, Giannantoni A, Massoud R, Dolci S, Micali F. Electromotive delivery of mitomycin C into human bladder wall. Cancer Res. 1997 Mar 1;57(5):875-80. PMID 9041189
- [Result] Di Stasi SM, Giannantoni A, Massoud R, Dolci S, Navarra P, Vespasiani G, Stephen RL. Electromotive versus passive diffusion of mitomycin C into human bladder wall: concentration-depth profiles studies. Cancer Res. 1999 Oct 1;59(19):4912-8. PMID 10519404
- [Result] Di Stasi SM, Giannantoni A, Stephen RL, Capelli G, Navarra P, Massoud R, Vespasiani G. Intravesical electromotive mitomycin C versus passive transport mitomycin C for high risk superficial bladder cancer: a prospective randomized study. J Urol. 2003 Sep;170(3):777-82. doi: 10.1097/01.ju.0000080568.91703.18. PMID 12913696
- [Result] Di Stasi SM, Giannantoni A, Giurioli A, Valenti M, Zampa G, Storti L, Attisani F, De Carolis A, Capelli G, Vespasiani G, Stephen RL. Sequential BCG and electromotive mitomycin versus BCG alone for high-risk superficial bladder cancer: a randomised controlled trial. Lancet Oncol. 2006 Jan;7(1):43-51. doi: 10.1016/S1470-2045(05)70472-1. PMID 16389183
- [Result] Di Stasi SM, Valenti M, Verri C, Liberati E, Giurioli A, Leprini G, Masedu F, Ricci AR, Micali F, Vespasiani G. Electromotive instillation of mitomycin immediately before transurethral resection for patients with primary urothelial non-muscle invasive bladder cancer: a randomised controlled trial. Lancet Oncol. 2011 Sep;12(9):871-9. doi: 10.1016/S1470-2045(11)70190-5. Epub 2011 Aug 8. PMID 21831711